CLINICAL TRIAL: NCT00334711
Title: A Prospective Study of Sulfonylureas in Patients With Diabetes Due to Kir6.2 Mutations
Brief Title: Sulfonylurea Response in Patients With Diabetes Due to Kir6.2 Mutations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Wellcome Trust (Other); Hôpital Necker-Enfants Malades (Other); Haukeland University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/10/196; 97/29/AH/mbs NTNU; Jnr 207/mkd NTNU; CCPPRB Necker GLIDKIR6.2
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-06

CONDITIONS: Diabetes Mellitus
Keywords: Permanent Neonatal Diabetes; Kir6.2; KCNJ11; Infancy onset diabetes; Sulfonylurea
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sulfonylurea Compounds

INTERVENTIONS:
Drug: Sulfonylurea

SUMMARY:
The purpose of this study is to investigate whether patients with diabetes due to Kir6.2 mutations can be treated with sulfonylurea medication rather than insulin, and if this is the case to investigate the mechanism for sulfonylurea response.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes due to KCNJ11 (Kir6.2) mutation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-01; Study Completion 2006-01

PRIMARY OUTCOMES:
HbA1c reduction

SECONDARY OUTCOMES:
insulin secretory response to intravenous glucose
insulin secretory response to oral glucose
insulin secretory response to mixed meal (sustacal)
Incidence of Hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, Study Director — Peninsula Medical School, Exeter, UK; Ewan R Pearson, Principal Investigator — Peninsula Medical School, Exeter, UK

REFERENCES:
- [Background] Gloyn AL, Pearson ER, Antcliff JF, Proks P, Bruining GJ, Slingerland AS, Howard N, Srinivasan S, Silva JM, Molnes J, Edghill EL, Frayling TM, Temple IK, Mackay D, Shield JP, Sumnik Z, van Rhijn A, Wales JK, Clark P, Gorman S, Aisenberg J, Ellard S, Njolstad PR, Ashcroft FM, Hattersley AT. Activating mutations in the gene encoding the ATP-sensitive potassium-channel subunit Kir6.2 and permanent neonatal diabetes. N Engl J Med. 2004 Apr 29;350(18):1838-49. doi: 10.1056/NEJMoa032922. PMID 15115830
- [Result] Pearson ER, Flechtner I, Njolstad PR, Malecki MT, Flanagan SE, Larkin B, Ashcroft FM, Klimes I, Codner E, Iotova V, Slingerland AS, Shield J, Robert JJ, Holst JJ, Clark PM, Ellard S, Sovik O, Polak M, Hattersley AT; Neonatal Diabetes International Collaborative Group. Switching from insulin to oral sulfonylureas in patients with diabetes due to Kir6.2 mutations. N Engl J Med. 2006 Aug 3;355(5):467-77. doi: 10.1056/NEJMoa061759. PMID 16885550
- See also: Related Info — http://www.diabetesgenes.org